CLINICAL TRIAL: NCT01066845
Title: Safety and Effectiveness of Adcirca (Tadalafil) in Japanese Patients With Pulmonary Arterial Hypertension: Open-label, Non-interventional Observational Study in Japan
Brief Title: Post Marketing Observational Study in Patients With Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 13693; H6D-JE-TD01 (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-02-03; First posted 2010-02-10 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Tadalafil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed Adcirca: all patients prescribed Adcirca during study period
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — prescribed in accordance with usual clinical practice
  Other Names: LY450190; Adcirca; Cialis

SUMMARY:
To investigate the long-term safety and effectiveness of Adcirca (tadalafil) in Pulmonary Arterial Hypertension (PAH) patients in the clinical practice -focused topics-

1. To evaluate the incidence of adverse events for the patients with long-term use
2. To evaluate the incidence of adverse events of decreased blood pressure, bleeding (including uterine hemorrhage), visual disturbance and sudden hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PAH receiving Adcirca

Exclusion Criteria:Patients who meet the criteria of contraindication

* patients with hypersensitivity to tadalafil
* patients who are using any form of organic nitrate
* patients with severe renal impairment
* patients with severe hepatic impairment
* patients taking strong inhibitors of CYP3A4
* patients taking strong inducers of CYP3A4

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients prescribed Adcirca from clinical practices
Sampling Method: Non-Probability Sample
Enrollment: 1809 (Actual)
Dates: Start 2010-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events related to decreased blood pressure, bleeding, visual disturbance and sudden hearing loss. | 2 years

SECONDARY OUTCOMES:
6 minute walk distance change from baseline | 2 years
World Health Organization (WHO) functional class change from baseline | 2 years
Survival time | 2 years
Pulmonary arterial pressure change from baseline | 2 years
Score change of Euro Quality of Life (EQ-5D) from baseline | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company